CLINICAL TRIAL: NCT04059861
Title: Ultrasound in Oral Tongue Cancer- Measurement of Depth of Invasion and Intraoperative Help in the Resection
Brief Title: Ultrasound in Tongue Cancer- a Help to Decide Depth of Invasion and to Improve the Surgical Margin
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Region Örebro County (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 252891
Record Dates: First submitted 2019-08-08; First posted 2019-08-16 (Actual); Last update posted 2021-12-27 (Actual); Status verified 2021-03

CONDITIONS: Tongue Cancer; Floor of Mouth Squamous Cell Carcinoma
Keywords: ultrasound; depth of invasion; tongue cancer; floor of the mouth cancer; resection margin; thickness; tongue carcinoma; tongue neoplasm; cancer of the tongue
MeSH Terms: conditions — Tongue Neoplasms; Margins of Excision | interventions — Ultrasonography

STUDY DESIGN:
Intervention Model Description: Clinical trial
Masking Description: The ultrasound examiner should not be aware of the results of the MRI.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ultrasound assisted resection (Other): resection of tongue cancer will be done with assistance of ultrasound to visualise the deep margin.
  Interventions: Diagnostic Test: Ultrasound

INTERVENTIONS:
Diagnostic Test: Ultrasound — enrolled patients will be investigated by ultrasound two times, awake in the clinic and in narcosis before the surgery. For those with tongue cancer ultrasound will be used during the surgery to visualise the deep margin of the tumour.

SUMMARY:
The purpose of this study is to investigate if ultrasound can be helpful in the diagnostic work-up of oral tongue and floor of the mouth cancer. One important factor is how deeply the tumour invades the tissue, the so called depth of invasion (DOI). The investigator will measure DOI with ultrasound and compare the result with the same measurement by magnetic resonance imaging and the microscopic result after the surgery (PAD).

Ultrasound will also be used during surgery of the tumour to investigate if it is useful to better decide the depth of the tumour and thereby improving the operation.

DETAILED DESCRIPTION:
The first part of this study will try to answer if ultrasound can improve the preoperative measurement of depth of invasion in tongue cancer and floor of the mouth cancer. The study population is new patients meeting the eligibility criteria presented to the hospital for treatment. Participants will be enrolled only after accepting the oral and written information and signing the written consent paper.

The examiner, one of three otorhinolaryngologists experienced in ultrasound, should be masked to the results of MRI. The first measurement is depth of invasion as well as thickness of the tumour in mm by palpation on awake patient. Thereafter the same measurements by ultrasound (BK Medical Medical flex focus 500, 18Mhz) with gel and protective cover is made with 0,5mm accuracy. Anesthetic gel or lingual block with carbocaine/adrenaline are provided as needed.

At the time of surgery the measurements above are done again on the patient in narcosis before the resection.

Images of the ultrasound measurements are saved for documentation. The results are compared to the corresponding measurements on MRI and also on PAD from the surgical specimen. PAD is considered gold standard.

Power calculation with help of biostatistician yielded a sample size of 55 patients, using a paired test with a 0,050 one-sided significance level will have 80% power to reject the null hypothesis that the proportions are not equivalent.

Analysis if ultrasound correctly classify the tumour´s DOI according to the TNM-classification 8th edition (<5mm, >5mm<10mm, >10mm) will be made.

The second part of the study will investigate if ultrasound during the surgical procedure can improve the discrimination of the deep margin of the tumour and thereby increasing the chance better surgical margins. The mucosal margins are marked in the usual fashion and the resection begins. After one fourth of the resection has been made, ultrasound is used to check that the deep margin is at least 10mm. This is repeated after one half and three quarters of the resection. At the end of the surgery a final ultrasound examination is made on the surgical specimen.

The margins obtained on PAD from resections done with ultrasound are compared to a matched retrospective group where the surgery was done without ultrasound.

After inclusion started our group started cooperation with another biostatician whom judged the analysis better be done from the quantitative variable of DOI in millimeter. This meant the power analysis shifted and a study population of between 15-23 participants was considered sufficient. Since the original plan was 55 participants we kept that number but after an interim analysis in may 2021 a total of 42 participants is now what we consider relevant in the study of DOI.

In our second endpoint studying ultrasound and surgical margin the interim analysis concluded that collection of patients for 2 years (may 2019 until may 2021) will be compared to a historical control group 4 years back in time (may 2015 until may 2019) and therefore the inclusion of that data stopped in may 2019.

ELIGIBILITY:
Inclusion Criteria:

biopsy verified tongue cancer or floor of the mouth cancer. International Statistical Classification of Diseases and Related Health Problems (ICD) 10 C02.0-2 or C04.0-1

Exclusion Criteria:

* former surgery in the oral cavity
* former radiation to the oral cavity
* floor of the mouth cancer not available to ultrasound investigation
* floor of the mouth cancer extending to the gingiva
* patients not suitable for surgery
* T4 tumours according to TNM 8
* age under 18
* patients declining to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2019-05-28 (Actual); Primary Completion 2021-11-29 (Actual); Study Completion 2021-11-29 (Actual)

PRIMARY OUTCOMES:
Depth of invasion | up to 6 weeks.
  Depth of invasion in millimeters measured by ultrasound compared to Clinical palpation , MRI and PAD.
Intraoperative ultrasound helpful during surgery | up to 6 weeks.
  Comparison of surgical margins in resections done with and without the assistance of ultrasound.

CONTACTS AND LOCATIONS:
Overall Officials: Johan Knutsson, Assoc. Prof., Principal Investigator — Region Örebro County
Locations (1):
- Örebro University Hospital, Örebro, Sweden

IPD SHARING:
Plan to Share IPD: Yes
The data of measurements will be shared.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 6 months after publication.
Access Criteria: Coded, computerized IPD will be available upon a request with the serious intention to improve the scientific knowledge and transparency.

REFERENCES:
- [Background] Baek CH, Son YI, Jeong HS, Chung MK, Park KN, Ko YH, Kim HJ. Intraoral sonography-assisted resection of T1-2 tongue cancer for adequate deep resection. Otolaryngol Head Neck Surg. 2008 Dec;139(6):805-10. doi: 10.1016/j.otohns.2008.09.017. PMID 19041507
- [Background] Kodama M, Khanal A, Habu M, Iwanaga K, Yoshioka I, Tanaka T, Morimoto Y, Tominaga K. Ultrasonography for intraoperative determination of tumor thickness and resection margin in tongue carcinomas. J Oral Maxillofac Surg. 2010 Aug;68(8):1746-52. doi: 10.1016/j.joms.2009.07.110. Epub 2009 Dec 23. PMID 20031291
- [Background] Tarabichi O, Kanumuri V, Juliano AF, Faquin WC, Cunnane ME, Varvares MA. Intraoperative Ultrasound in Oral Tongue Cancer Resection: Feasibility Study and Early Outcomes. Otolaryngol Head Neck Surg. 2018 Apr;158(4):645-648. doi: 10.1177/0194599817742856. Epub 2017 Nov 21. PMID 29161194
- [Background] Lydiatt WM, Patel SG, O'Sullivan B, Brandwein MS, Ridge JA, Migliacci JC, Loomis AM, Shah JP. Head and Neck cancers-major changes in the American Joint Committee on cancer eighth edition cancer staging manual. CA Cancer J Clin. 2017 Mar;67(2):122-137. doi: 10.3322/caac.21389. Epub 2017 Jan 27. PMID 28128848
- [Background] International Consortium for Outcome Research (ICOR) in Head and Neck Cancer; Ebrahimi A, Gil Z, Amit M, Yen TC, Liao CT, Chaturvedi P, Agarwal JP, Kowalski LP, Kreppel M, Cernea CR, Brandao J, Bachar G, Bolzoni Villaret A, Fliss D, Fridman E, Robbins KT, Shah JP, Patel SG, Clark JR. Primary tumor staging for oral cancer and a proposed modification incorporating depth of invasion: an international multicenter retrospective study. JAMA Otolaryngol Head Neck Surg. 2014 Dec;140(12):1138-48. doi: 10.1001/jamaoto.2014.1548. PMID 25075712
- [Background] Lam P, Au-Yeung KM, Cheng PW, Wei WI, Yuen AP, Trendell-Smith N, Li JH, Li R. Correlating MRI and histologic tumor thickness in the assessment of oral tongue cancer. AJR Am J Roentgenol. 2004 Mar;182(3):803-8. doi: 10.2214/ajr.182.3.1820803. PMID 14975989
- [Background] Yesuratnam A, Wiesenfeld D, Tsui A, Iseli TA, Hoorn SV, Ang MT, Guiney A, Phal PM. Preoperative evaluation of oral tongue squamous cell carcinoma with intraoral ultrasound and magnetic resonance imaging-comparison with histopathological tumour thickness and accuracy in guiding patient management. Int J Oral Maxillofac Surg. 2014 Jul;43(7):787-94. doi: 10.1016/j.ijom.2013.12.009. Epub 2014 Mar 2. PMID 24598430
- [Background] Alsaffar HA, Goldstein DP, King EV, de Almeida JR, Brown DH, Gilbert RW, Gullane PJ, Espin-Garcia O, Xu W, Irish JC. Correlation between clinical and MRI assessment of depth of invasion in oral tongue squamous cell carcinoma. J Otolaryngol Head Neck Surg. 2016 Nov 22;45(1):61. doi: 10.1186/s40463-016-0172-0. PMID 27876067
- [Background] Klein Nulent TJW, Noorlag R, Van Cann EM, Pameijer FA, Willems SM, Yesuratnam A, Rosenberg AJWP, de Bree R, van Es RJJ. Intraoral ultrasonography to measure tumor thickness of oral cancer: A systematic review and meta-analysis. Oral Oncol. 2018 Feb;77:29-36. doi: 10.1016/j.oraloncology.2017.12.007. Epub 2017 Dec 18. PMID 29362123
- [Derived] Nilsson O, Knutsson J, Landstrom FJ, Magnuson A, von Beckerath M. Ultrasound-assisted resection of oral tongue cancer. Acta Otolaryngol. 2022 Sep-Dec;142(9-12):743-748. doi: 10.1080/00016489.2022.2153916. Epub 2022 Dec 20. PMID 36537851